CLINICAL TRIAL: NCT04613544
Title: A Prospective, Open Label, Multi-Center, Pilot Study to Assess Safety, Efficacy and Usability of Application for Atrial Fibrillation Vocal Marker
Brief Title: Assess Safety, Efficacy and Usability of Application for Atrial Fibrillation Vocal Marker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiokol Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-120
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Atrial fibrillation diagnosed patients.
  Interventions: Device: Voice Assist Arrhythmia Monitoring (VAAM)

INTERVENTIONS:
Device: Voice Assist Arrhythmia Monitoring (VAAM) — application flag the potential occurrence of irregular heart rhythms suggestive of atrial fibrillation (AF) and notify to further investigate the occurrence of the suspected AF episode by prompting user to initiate ECG test to confirm.

SUMMARY:
Voice Assist Arrhythmia Monitoring (VAAM) is an application running on smartphones and/or landline phones that performs vocal tests for the monitoring of abnormalities in the heart rhythm.

DETAILED DESCRIPTION:
Following ICF signature and process and eligibility confirmation, subject will have a training session to assure correct application use. The subjects will be asked to pronounce few vowels 3 times a day to be evaluated by the application analysis algorithm at the patient natural environment.

At the same time, a single lead ECG system will be recorded synchronously ECG for reference with the use of dedicated recording device

ELIGIBILITY:
Inclusion Criteria:

1. Female and male at age of ≥18 years and above.
2. All AF types Or Medical history of Cryptogenic stroke.
3. Ability and willingness to sign an informed consent form

Exclusion Criteria:

1. Subjects with implanted cardiac defibrillators or pacemakers neurostimulators and/or body worn medical devices such as insulin pumps.
2. Subjects diagnosed with any heart arrhythmias other than A-Fib, except for PVC.
3. Patient who underwent cardioversion or ablation in the last year and is in stable sinus rhythm.
4. Women who are pregnant or breastfeeding (women of child-bearing potential must provide a declaration stating that they are not pregnant)
5. Tremor or Parkinson's disease
6. Current hoarseness
7. Barriers for communication and lack of capability to execute the handlings required for this study.
8. Subjects who are currently enrolled in another clinical investigation. Parallel Enrollment to a non-interventional study is permitted.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial Fibrillation Diagnosed
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | 6 weeks
  related Adverse device effect

SECONDARY OUTCOMES:
Usability | 6 weeks
  Assessment of User Experience and User Interface
Effectivness | 6 wweeks
  application specificity and sensitivity

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva